CLINICAL TRIAL: NCT01803256
Title: The Measurement of Spine Dynamics During Gait for the Quantification of Intervention Outcomes in Patients With Different Pathologies
Brief Title: Possibilities and Limitations of a New Method for the Measurement of Spine Dynamics During Gait
Status: Completed | Type: Observational
Sponsor: University Children's Hospital Basel (Other)
Collaborators: Swiss Federal Institute of Technology (Other); Bern University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Prof. Reinald Brunner, MD, Doctor in Charge, Neuro-Orthopedics, University Children's Hospital Basel
Other Study IDs: UKBB-Spine-1315-1
Record Dates: First submitted 2013-02-26; First posted 2013-03-04 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Scoliosis patients:: 15 patients with adolescent idiopathic scoliosis.
- Control subjects:: 15 adolescent healthy control subjects

SUMMARY:
The full body marker sets that are typically used in opto-electronic 3D gait analyses either disregard the spine entirely or regard it as a rigid structure. Therefore, the purpose of this study is to identify the possibilities and limitations of an enhanced trunk marker set for the measurement of spine dynamics during gait in adolescents with and without structural spine deformities.

It has been hypothesized that the enhance trunk marker set:

1. is a valid method for the measurement of spine deformations in the sagittal, frontal and indirectly transverse planes.
2. is an applicable and reliable method for the measurement of spine dynamics during gait in healthy adolescents and in patients with structural deformities such as seen in scoliosis.
3. is sensitive enough to distinguish the spinal movement pattern during gait measured in scoliosis patients from the one measured in healthy adolescents.

To verify the hypotheses, the following measurements will be carried out:

* Biplanar radiographs (a-p and lateral) with radio-opaque markers in scoliosis patients.
* Instrumented gait analysis with a standard full body marker set and the enhanced trunk marker set in scoliosis patients and healthy controls.

ELIGIBILITY:
Scoliosis patients:

Inclusion Criteria:

* Adolescent idiopathic scoliosis
* Able to walk a distance of minimum 50 meters barefoot and without any assistive device

Exclusion Criteria:

* Other types of scoliosis (e.g. of neurological origin)
* Previous treatment of scoliosis (conservative or surgery)
* Injuries of the locomotor system which led to persistent deformities

Healthy controls:

Exclusion Criteria:

* Any pathologies or diseases affecting the locomotor system
* Injuries to the locomotor system which led to persistent deformities
* Obesity (> 95th BMI-per-age percentile)
* Leg length discrepancy (more than 1% of body height)

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Scoliosis patients: Patients attending the Orthopedic Department at UKBB for scoliosis treatment.
  Healthy controls: Middle and high school students in the Basel area.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-04; Primary Completion 2014-09 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Validity of the enhanced trunk marker set for a static measurement of spinal kinematics (radiographic vs. motion analysis measurements). | Data will be collected between April 2013 and June 2014. For each scoliosis patient, the radiographic measurements will be conducted immediately after inclusion and the motion analysis measurements within 48 hours of the radiographic measurements.
  This primary endpoint will only be evaluated in scoliosis patients since healthy adolescents do not undergo radiographic measurements. Parameters include lumbar and thoracic spine curvature angles in the sagittal and frontal planes.
Reliability of the enhanced trunk marker set for the measurement of spinal kinematics in scoliosis patients and healthy adolescents during gait. | Data will be collected between April 2013 and June 2014. Spinal kinematics during gait will be measured in each scoliosis patient / healthy adolescent within 48 hours of the radiographic examination.
  Parameters include lumbar, thoracic and cervical spine curvature angles in the sagittal and frontal planes and segmental rotation angles in the transverse plane.
Differences in spinal kinematics between scoliosis patients and healthy adolescents during gait. | Data will be collected between April 2013 and June 2014. Spinal kinematics during gait will be measured in each scoliosis patient / healthy adolescent within 48 hours of the radiographic examination.
  Parameters include lumbar, thoracic and cervical spine curvature angles in the sagittal and frontal planes and segmental rotation angles in the transverse plane.

SECONDARY OUTCOMES:
Differences in spatio-temporal gait parameters and kinematics and kinetics of peripheral joints between scoliosis patients and healthy adolescents during gait. | Data will be collected between April 2013 and June 2014. Parameters during gait will be measured in each scoliosis patient / healthy adolescent within 48 hours of the radiographic examination.
  Parameters include gait speed, cadence and single and double limb support as well as angles, torques and powers of peripheral joints in all three planes.

CONTACTS AND LOCATIONS:
Overall Officials: Reinald Brunner, MD, Principal Investigator — University Children's Hospital Basel; Stefan Schmid, PT, PhD, Study Chair — Swiss Federal Institute of Technology / Bern University of Applied Sciences; Silvio Lorenzetti, PhD, DSc, Study Director — Swiss Federal Institute of Technology; Jacqueline Romkes, PhD, Study Director — University Children's Hospital Basel; Carol-Claudius Hasler, MD, Study Director — University Children's Hospital Basel
Locations (1):
- University Children's Hospital Basel, Basel, Switzerland

REFERENCES:
- [Result] Schmid S, Studer D, Hasler CC, Romkes J, Taylor WR, Brunner R, Lorenzetti S. Using Skin Markers for Spinal Curvature Quantification in Main Thoracic Adolescent Idiopathic Scoliosis: An Explorative Radiographic Study. PLoS One. 2015 Aug 13;10(8):e0135689. doi: 10.1371/journal.pone.0135689. eCollection 2015. PMID 26270557
- [Result] Schmid S, Studer D, Hasler CC, Romkes J, Taylor WR, Lorenzetti S, Brunner R. Quantifying spinal gait kinematics using an enhanced optical motion capture approach in adolescent idiopathic scoliosis. Gait Posture. 2016 Feb;44:231-7. doi: 10.1016/j.gaitpost.2015.12.036. Epub 2015 Dec 29. PMID 27004664